CLINICAL TRIAL: NCT05635968
Title: The Multicenter Phase II Clinical Trial for Evaluation of Safety and Efficacy Using Low Dose Irradiation With Alzheimer's Disease
Brief Title: The Clinical Trial of Low Dose Irradiation for Alzheimer's Disease
Acronym: LDRT-AD-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Collaborators: Korea Hydro&Nuclear Power Radiation Health Institute (Unknown); Chungbuk National University Hospital (Other); SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Weon Kuu Chung, Professor, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KHNMC 2022-03-030
Record Dates: First submitted 2022-10-28; First posted 2022-12-02 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
Keywords: radiation therapy; Low-dose whole brain irradiation
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: single blinded (subject)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-dose whole brain irradiation group 1 (4cGy/day) (Experimental): Low-dose whole brain irradiation with general AD medication treatment (4cGy/day, 2times/1wk, total 24cGy, 6 times/3wks)
  Interventions: Radiation: Low-dose whole brain irradiation
- Low-dose whole brain irradiation group 2 (50cGy/day) (Experimental): Low-dose whole brain irradiation with general AD medication treatment (50cGy/day, 2times/1wk, total 300cGy, 6 times/3wks)
  Interventions: Radiation: Low-dose whole brain irradiation
- Sham RT group (Sham Comparator): Sham RT wtih general AD medication treatment (0cGy/day, 2times/1wk, total 0cGy, 6 times/3wks)
  Interventions: Radiation: Low-dose whole brain irradiation

INTERVENTIONS:
Radiation: Low-dose whole brain irradiation — In the experimental group (1), 20 patients receive 4cGy x 6 times, a total of 24 cGy of irradiation. In the experimental group (2), 20 patients receive 50 cGy x 6 times, a total of 300 cGy of irradiation. All experimental groups and control group visit the hospital about 1, 6, and 12 months after irradiation to evaluate efficacy and safety.

SUMMARY:
This is a phase II, multicenter, prospective, randomized controlled trial to treat patients with Alzheimer's disease (AD) using low-dose irradiation (LDIR). This study aims to evaluate the safety and efficacy of LDIR to whole brain in patients with AD and to determine the potentially applicable radiation dose.

DETAILED DESCRIPTION:
Screening tests, cognitive function tests, brain MRI, and amyloid PET are performed on subjects who voluntarily consent in writing to participate in the trial to determine whether they meet the inclusion/exclusion criteria. Randomization is assigned to eligible subjects. The experimental groups are irradiated six times for 3 weeks according to the radiation dose determined for each group, and the control group is irradiated with sham radiation. The patients assigned to the experimental group receive whole brain irradiation with 6 MV energy using a linear accelerator. In the experimental group (1), 20 patients receive 4cGy x 6 times, a total of 24 cGy of irradiation. In the experimental group (2), 20 patients receive 50 cGy x 6 times, a total of 300 cGy of irradiation. All experimental groups and control group visit the hospital about 1, 6, and 12 months after irradiation to evaluate efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria are satisfied for the subjects to be included in the study:

1. Aged between 60 and 85 years.
2. Diagnosed with probable Alzheimer's disease (AD) dementia based on the new diagnostic criteria for Alzheimer's disease outlined by the National Institute on Aging and Alzheimer's Association (NIA-AA).
3. Stably maintaining the general AD drug treatment (donepezil, galantamine, rivastigmine, or memantine) for more than 3 months.
4. Amyloid accumulation in brain confirmed by Amyloid PET.
5. Mild AD (score range of 13 to 24 on the Korean Mini-Mental State Examination (K-MMSE) or 0.5 or 1 on the Clinical Dementia Rating scale (CDR)).
6. Able to perform cognitive function tests and imaging tests.
7. Accompanied by a guardian who provides information on the subject's overall status, cognitive function, and functional changes.
8. Written informed consent was provided by the subject or the guardian to participate in this trial.

Exclusion Criteria:

Subjects who fall under any of the following criteria are excluded from the study:

1. Previous history of radiation to the brain.
2. History of seizure within the previous 10 years of the screening time.
3. Skin disease on the scalp.
4. Previous history of malignancy.
5. Pregnancy or breastfeeding.
6. Subjects with cognitive decline associated with drugs or neurological / neurodegenerative conditions, not AD (i.e., drug abuse, vitamin B12 deficiency, thyroid dysfunction, stroke or other cerebrovascular conditions, Lewy body dementia, frontotemporal dementia, and head trauma).
7. Clinically significant, unstable mental illness (i.e., uncontrolled depression, schizophrenia, and bipolar disorder) within the last 6 months.
8. Subjects whose brain MRI confirms evidence of: acute or subacute hemorrhage, prior macro hemorrhage (defined as >1 cm in diameter, T2 sequence) or prior subarachnoid hemorrhage unless it can be documented that the finding is not due to an underlying structural or vascular abnormality, more than 4 microhemorrhages, cortical infarct (defined as >1.5 cm in diameter, irrespective of anatomic location), >1 lacunar infarct (defined as >1.5 cm in diameter), superficial siderosis, and history of diffuse white matter disease as defined by a score of 3 on the age-related white matter changes scale. Any finding that, in the opinion of the investigator, might be a contributing cause of the subject's dementia, or pose a risk to the subject, or might prevent a satisfactory MRI assessment for safety monitoring are also included in the exclusion criteria.
9. Those who have other findings that are considered clinically important, and those who are judged by the researcher to be inappropriate for participation in this study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
saftey and efficacy | 6 months after completion of low-dose irradiation to whole brain
  1) Changes in cognitive function test score compared to baseline after six months are estimated using Alzheimer's disease assessment scale-Korea (ADAS-K) (range 0-70, higher scrores mean a worse outcome). The amount of change is evaluated as a valid response if it shows an improvement of 5% or more compared to the baseline score.
saftey and efficacy | 6 months after completion of low-dose irradiation to whole brain
  2) Number of adverse events 6 months after baseline determined by the Radiation Therapy Oncology Group (RTOG) toxicity grading system.

SECONDARY OUTCOMES:
Changes in cognitive function test score | 6 months after completion of low-dose irradiation to whole brain
  If the cognitive function test such as Korean-Mini-Mental Status Examination (K-MMSE)(range 0-30, higher scrores mean a better outcome) showed an improvement of 5% or more after six months, it was evaluated as an effective response.
Changes in cognitive function test score | 6 months after completion of low-dose irradiation to whole brain
  If the cognitive function test such as Clinical Dementia Rating scale (CDR)(range 0-3, higher scrores mean a worse outcome) showed an improvement of 5% or more after six months, it was evaluated as an effective response.
Changes in cognitive function test score | 6 months after completion of low-dose irradiation to whole brain
  If the cognitive function test such as Caregiver Administered-Neuropsychiatric Inventory (CGA-NPI)(range 0-144, higher scrores mean a worse outcome) showed an improvement of 5% or more after six months, it was evaluated as an effective response.
Changes in cognitive function test score | 6 months after completion of low-dose irradiation to whole brain
  If the cognitive function test such as Korean Intstrumental Activities of Daily Living (K-iADL)(range 10-33, higher scrores mean a worse outcome) showed an improvement of 5% or more after six months, it was evaluated as an effective response.
Changes in the standardized uptake value ratio (SUVR) | 6 months after completion of low-dose irradiation to whole brain
  Changes in the standardized uptake value ratio (SUVR) of the amyloid PET in the frontal, parietal, lateral temporal, anterior wedge lobe, and the posterior gyrus are evaluated. It was considered as an effective response if the change of SUVR shows an improvement of 5% or more 6 months after the completion of LDIR.

CONTACTS AND LOCATIONS:
Overall Officials: Weon-Kuu Chung, MD, PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim DY, Kim JS, Seo YS, Park WY, Kim BH, Hong EH, Kim JY, Cho SJ, Rhee HY, Kim A, Kim KY, Oh DJ, Chung WK. Evaluation of Efficacy and Safety Using Low Dose Radiation Therapy with Alzheimer's Disease: A Protocol for Multicenter Phase II Clinical Trial. J Alzheimers Dis. 2023;95(3):1263-1272. doi: 10.3233/JAD-230241. PMID 37638435